CLINICAL TRIAL: NCT05881096
Title: Effectiveness of START (Startle Adjuvant Rehabilitation Therapy) in Enhancing Upper Extremity Function Post-Stroke
Brief Title: Effectiveness of START (Startle Adjuvant Rehabilitation Therapy) in Enhancing Arm Function Post-Stroke
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Claire Honeycutt, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002440b
Record Dates: First submitted 2023-02-21; First posted 2023-05-31 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: Hemiplegia; Upper extremity impairment
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- START (Startle Adjuvant Rehabilitation Therapy) (Experimental): Participants in this group practice a functional reaching task with the START condition (startling acoustic stimuli applied during 33% of trials).
  Interventions: Other: START - Startle Adjuvant Rehabilitation Therapy
- Control (Sham Comparator): Participants in this group will practice a functional reaching task without the START (Startle Adjuvant Rehabilitation Therapy) intervention
  Interventions: Other: Sham Control

INTERVENTIONS:
Other: START - Startle Adjuvant Rehabilitation Therapy — Application of startling acoustic stimuli during practice of movement task
  Arms: START (Startle Adjuvant Rehabilitation Therapy)
Other: Sham Control — Practice of movement task without START
  Arms: Control

SUMMARY:
The goal of this clinical trial is to test the effectiveness of START (Startle Adjuvant Rehabilitation Therapy) in improving arm function after a stroke. The main questions it aims to answer are 1) Does startle rehabilitation therapy improve functional arm performance after training on a specific task and 2) Can training benefits, if any, be seen in other untrained tasks? Researchers will enroll participants across a wide range of upper extremity impairments post-stroke. Participants will be enrolled in three consecutive days of in-person training on an upper extremity task followed by a single-day follow-up session one month after training is completed. Each training session will last for approximately 3 hours per day. Participants will be randomly assigned to one of two groups; 1) Arm training with START and 2) Arm training without START. Study participants and assessors will be blinded to the type of training received. Before the training, participants will be clinically assessed to determine impairment level. During training, participants will be asked to perform; 1) a simulated feed task which involves transferring kidney beans using a spoon from one cup (start position) to another cup (end position) in front of them OR 2) A functional reaching task where participants will maintain a tool (spoon) in their hand while extending their arm forward towards an end position based on the severity of arm impairment as determined by the clinical assessment. Researchers will compare the % change in trained task scores, muscle activity, and arm movement outcome measures at three-time points; baseline on day 1, at the end of training on day 3, and one month after training.

DETAILED DESCRIPTION:
A patient's socioeconomic status (SES) should not predict their post-stroke disability but individuals with low SES are more disabled and have higher mortality rates compared to individuals with high SES. These inequities are not isolated to low- and middle-income countries. In the United States, individuals with low SES are more disabled at 3 months and less likely to be independently ambulatory or discharged to their own homes. There are many factors contributing to these outcomes; however, one critical feature is access to affordable care. Many newly developed rehabilitation therapies and technologies require expensive equipment (e.g. instrumented treadmills, transcranial magnetic stimulation) and extensive training for clinical staff. The extra costs (financial and training) ensure that these state-of-the-art options are only available at metropolitan, well-funded institutions or to individuals who can afford additional healthcare costs. There is an urgent need for accessible, low-cost solutions capable of being delivered at underfunded hospitals and to individuals with no or low insurance coverage.

Startle Adjuvant Rehabilitation Therapy (START) represents an accessible and low-cost solution that can be delivered to rural and socioeconomically disadvantaged populations. START is the application of a startling, acoustic stimulus alongside traditional therapy. Distinct from other auditory treatments (e.g. metronome, music), administration of a START represents an endogenous activation of the brainstem (i.e. reticular formation) a phenomenon referred to as startReact. Rather than being a standalone treatment, START is adjuvant. An adjuvant is considered the introduction of an agent (traditionally pharmacological) that contributes to or enhances an existing medical regimen. Similarly, START is applied within a standard clinical practice to enhance and accelerate skill re-learning through activation of the brainstem.

START has been advanced as an adjuvant therapy tool because of the profound way it enhances training outcomes in individuals with stroke, in particular severe stroke. This is particularly compelling given the high degree of difficulty in generating functional changes in individuals with chronic, severe stroke. There is emerging evidence that individuals with stroke strengthen ipsilateral reticulospinal connections during the process of recovery. Thus, START may represent a priming of the nervous system to engage the reticular formation, which is nearly always spared post-stroke, during therapy to enhance both training and long-term outcomes. Though provocative, there are critical gaps in the literature that are required before START can be deployed in the clinic. Here, the investigators propose to 1) perform a rigorous randomized controlled trial during tasks of functional significance (Aim 1), and 2) assess the capacity of START training to generalize to untrained tasks (Aim 2).

Aim 1: Evaluate the capacity of START to enhance training outcomes in individuals with stroke (iwS). The objective of this aim is to demonstrate that START can enhance tasks of clinical and functional significance like those performed during therapy. The investigators propose a randomized, single-blind, parallel, controlled trial evaluating the impact of START on training outcomes of a functional reaching task in iwS. Hypothesis 1: The rate of learning and retention will be larger during training with START compared to control (training without START).

Aim 2: Evaluate the generalizability of START training to untrained tasks. To be viable as an adjuvant clinical tool to enhance activities of daily living, training benefits attributable to START must translate beyond the specific tasks trained during therapy. The investigators propose to evaluate skill transference using sorting and dressing tasks. Hypothesis 2: Training with START will show higher skill transfer (e.g. time to complete sorting/dressing task) compared to training without START.

SIGNIFICANCE & IMPACT Imagine the transformative impact of an inexpensive tool that could be implemented not only in well-funded, metropolitan hospitals but also in small, rural, and socioeconomically disadvantaged hospitals enhancing recovery for iwS regardless of disability severity, socioeconomic status, or location. Every year, $43,000,000,000 is paid for care and therapy of the 7,000,000 stroke survivors living in the US but six months post-stroke 65% of patients cannot use their impaired hand during activities of daily living (e.g. feeding, toileting) and 63.5% of stroke survivors will never achieve a total Fugl-Meyer score greater than 90/226 - i.e. severe disability. These statistics are worse for individuals with low SES. A recent, 2018 study demonstrated that patients from low SES backgrounds received less in-patient and out-patient care and were discharged more quickly leading to higher levels of disability and mortality.

If successful, this study will revolutionize treatment for stroke survivors because START is non-invasive, inexpensive, and mobile making it accessible to rural and socioeconomically disadvantaged populations. START's application is a loud, acoustic stimulus timed with planned motor activity and can be administered via headphones. Unlike many new rehabilitation devices/techniques, START represents an extremely safe intervention (the application is a loud sound well beneath OSHA (Occupational Safety and Health Administration) regulations with no reported adverse reactions since its discovery. Thus, clinical staff training and safety protocols are minimal further decreasing application costs. Finally, it is mobile and easily packaged, so it can be administered via the increasing number of telemedicine programs designed for rural populations. Finally, START allows severe stroke survivors to participate in and benefit from therapy. The benefits of START are not contained to severe stroke survivors (e.g. improvement of hand extension in mildly disabled patients) but the capacity of START to work in severe patients significantly increases the potential of this tool to assist patients across all levels of disability.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Capacity to provide informed consent
3. Cerebral stroke at least 6 months prior to testing
4. Presence of severe-to-mild upper extremity impairment
5. Corrected pure tone threshold (octave frequencies 250- 4000 Hz) norms for their age and gender. NOTE: Audiometry data will be collected for all participants by lab personnel trained by an audiologist in a sound-attenuated booth. The investigators expect that ~30% of participants will use hearing aids; the investigators will not exclude these individuals but rather include hearing aid use as a covariate in analyses.

Exclusion Criteria:

1. Severe concurrent medical problems (e.g. uncontrolled cardiorespiratory impairment)
2. Acute/painful condition/injury of upper extremity/spine that interfere with ability to participate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in EMG (electromyography) onset (in ms) during functional reaching task | Change in EMG onset from baseline (before training on day 1) to post (after training on day 3)
  Evaluation of EMG onset measured in milliseconds (ms) for different muscles of the affected / most affected arm. EMG activity will be recorded using Ag/Cl surface electrodes and onset will be detected using a custom MATLAB code.
Change in EMG (electromyography) amplitude (in mV) during the functional reaching task | Change in EMG amplitude from baseline (before training on day 1) to post (after training on day 3)
  Evaluation of EMG amplitude measured in millivolts(mV) for different muscles of the affected / most affected arm. EMG activity will be recorded using Ag/Cl surface electrodes and amplitude will be detected using a custom MATLAB code.
Change in movement onset (in ms) on functional reaching task | Change in movement onset from baseline (before training on day 1) to post (after training on day 3)
  Evaluation of movement onset in milliseconds(ms). Movement activity will be measured using Infrared(IR) markers placed at fixed joint locations on the arm. Movement onset will be detected using a custom MATLAB code.
Change in movement linearity (in mm) on functional reaching task | Change in movement linearity from baseline (before training on day 1) to post (after training on day 3)
  Evaluation of movement linearity in millimeters (mm). Movement activity using Infrared(IR) markers placed at fixed joint locations on the arm. Movement linearity will be evaluated using a custom MATLAB code.
Change in functional reaching task scores during training | Change in functional reaching task scores from on day 1 of training compared to day 3 of training
  The functional reaching task (simulated feeding task) is scored based on the number of successful repetitions i.e. the total number of kidney beans successfully transferred or dropped.
Change in functional reaching task scores | Change in functional reaching task scores from baseline (before training on day 1) to post (after training on day 3)
  The functional reaching task (simulated feeding task) is scored based on the number of successful repetitions i.e. the total number of kidney beans successfully transferred or dropped.
Change in sorting task scores | Change in sorting task scores from baseline (before training on day 1) to post (after training on day 3)
  The change in sorting task scores will be used to evaluate skill transfer. The sorting evaluates an untrained task with spatiotemporally similar characteristics to the trained task. A higher score indicates a better performance.
Change in dressing task scores | Change in dressing task scores from baseline (before training on day 1) to post (after training on day 3)
  The change in dressing task scores will be used to evaluate skill transfer. The dressing task evaluates an untrained task with spatiotemporally dissimilar characteristics to the trained task. A higher score indicates a better performance.

SECONDARY OUTCOMES:
Retention in functional reaching task scores | Retention of functional reaching task comparing immediately after training on day 3 to one-month post
  Functional reaching task (Trained task - simulated feeding task). Functional reaching task scores is computed as the number of beans transferred and dropped within a given time frame.
Retention in skill transfer 1 : sorting task scores | Retention of sorting task comparing immediately after training on day 3 to one-month post
  sorting task (untrained task) scores will be calculated as the number of blocks successfully transferred. The higher the number of blocks transferred (higher score), the better the performance.
Retention in skill transfer 2: dressing task | Retention of sorting task comparing immediately after training on day 3 to one-month post
  dressing task (untrained task) scores will be computed as the number of buttons/velcro successfully fastened within a given time frame. The higher the score, the better the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States